CLINICAL TRIAL: NCT03236246
Title: Study of KRX-0502 (Ferric Citrate) Dose Regimens in Subjects With Non-Dialysis Dependent Chronic Kidney Disease and Iron-Deficiency Anemia
Brief Title: KRX-0502 (Ferric Citrate) in Subjects With NDD-CKD and IDA (The COMPASS Trial)
Acronym: COMPASS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Keryx Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KRX-0502-402
Record Dates: First submitted 2017-07-26; First posted 2017-08-01 (Actual); Results first posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Chronic Kidney Diseases; Iron Deficiency Anemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia, Iron-Deficiency | interventions — ferric citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): KRX-0502 1 tablet thrice daily (TID) with meals
  Interventions: Drug: KRX-0502
- Group 2 (Experimental): KRX-0502 2 tablets twice daily (BID) with the largest 2 daily meals
  Interventions: Drug: KRX-0502

INTERVENTIONS:
Drug: KRX-0502 — Oral ferric citrate with meals
  Other Names: ferric citrate

SUMMARY:
The objectives of this study are to assess the long-term efficacy and safety of different dose regimens of KRX-0502 in the treatment of iron deficiency anemia (IDA) in adult subjects with non-dialysis dependent chronic kidney disease (CKD).

DETAILED DESCRIPTION:
This is a Phase 4, 48-week, randomized, open-label, multicenter clinical study comprised of 2 periods: a 24-week Dose Titration Period, followed by a 24-week Dose Maintenance Period. The study will consist of 12 scheduled clinic visits over a period of 48 weeks and additional visits as needed.

ELIGIBILITY:
Inclusion Criteria:

* Estimated glomerular filtration rate ≥20 mL/min and <60 mL/min
* Hgb ≥8.5 g/dL and ≤11.5 g/dL
* Serum ferritin ≤500 ng/mL and transferrin saturation (TSAT) ≤25%
* Serum intact parathyroid hormone ≤600 pg/mL

Exclusion Criteria:

* Serum phosphate <3.0 mg/dL
* Intravenous (IV) iron administered within 4 weeks prior to Screening
* Erythropoiesis-stimulating agents (ESA) administered within 4 weeks prior to Screening
* Blood transfusion within 4 weeks prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Keryx Biopharmaceuticals
Locations (27):
- United States (27):
  - Arizona Kidney Disease and Hypertension center: AKDHC Medical Research Services, LLC, Phoenix, Arizona
  - California Institute of Renal Research, Chula Vista, California
  - California Institute of Renal Research, El Centro, California
  - California Institute of Renal Research, Poway, California
  - Denver Nephrologists, P.C., Denver, Colorado
  - Miami Kidney Group, Miami, Florida
  - Kidney and Hypertension Specialists of Miami, P.A., Miami, Florida
  - Southeastern Clinical Research Institute, LLC, Augusta, Georgia
  - Renal Associates, LLC, Columbus, Georgia
  - Research by Design, LLC, Chicago, Illinois
  - South Mississippi Medical Research, LLC, Gulfport, Mississippi
  - Clinical Research Consultants, Kansas City, Missouri
  - Sierra Nevada Nephrology Consultants, Reno, Nevada
  - Hypertension and Nephrology Association, Eatontown, New Jersey
  - Division of Kidney/HTN Research, Great Neck, New York
  - Mountain Kidney & Hypertension Associates, Asheville, North Carolina
  - Metrolina Nephrology Associates, PA, Charlotte, North Carolina
  - Eastern Nephrology Associates, Greenville, North Carolina
  - Southeastern Nephrology Associates, Jacksonville, North Carolina
  - Eastern Nephrology Associates, New Bern, North Carolina
  - Southeastern Nephrology, Wilmington, North Carolina
  - Columbia Nephrology Associates, PA, Columbia, South Carolina
  - South Carolina Nephrology & Hypertension Center, Inc, Orangeburg, South Carolina
  - Nephrology Associates, P.C., Nashville, Tennessee
  - Research Management, Inc., Austin, Texas
  - P & I Clinical Research, LLC, Lufkin, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- KRX-0502 3 g/Day: Participants were randomized to receive KRX-0502 3 grams per day (g/day), administered as 1 tablet 3 times daily (TID) (total of 3 tablets/day) with meals, in the 24-week Dose Titration Period. Scheduled study drug dose adjustment occurred at Week 12 and was based upon the hemoglobin (Hgb) increase relative to Baseline and an Hgb threshold. Participants who completed the 24-week Dose Titration Period were eligible to enter the 24-week Dose Maintenance Period. During the Dose Maintenance Period, participants continued on the dose determined during the Dose Titration Period. The maximum dose was the dose determined at Week 12.
- KRX-0502 4 g/Day: Participants were randomized to receive KRX-0502 4 g/day, administered as 2 tablets twice daily (BID) with the larger of 2 daily meals, in the 24-week Dose Titration Period. Scheduled study drug dose adjustment occurred at Week 12 and was based upon the Hgb increase relative to Baseline and an Hgb threshold. Participants who completed the 24-week Dose Titration Period were eligible to enter the 24-week Dose Maintenance Period. During the Dose Maintenance Period, participants continued on the dose determined during the Dose Titration Period. The maximum dose was the dose determined at Week 12.
Period: 24-Week Dose Titration Period
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Started | 104 | 102
Completed | 80 | 75
Not Completed | 24 | 27
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Lost to Follow-up | 0 | 2
Not completed — Study Drug Non-Compliance | 3 | 2
Not completed — Investigator Judgement | 1 | 1
Not completed — Prohibited Therapy | 1 | 1
Not completed — Start Chronic Dialysis/Kidney Transplant | 0 | 1
Not completed — Death | 3 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Adverse Event | 7 | 8
Not completed — Captured as Other | 1 | 2
Period: 24-Week Dose Maintenance Period
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Started | 76 (Not all participants completing the Dose Titration Period opted to enter the Dose Maintenance Period) | 72 (Not all participants completing the Dose Titration Period opted to enter the Dose Maintenance Period)
Completed | 73 | 66
Not Completed | 3 | 6
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Prohibited Therapy | 1 | 0
Not completed — Death | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who took at least 1 dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day | Total
Number analyzed (Participants) | 104 | 101 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (11.22) | 69.9 (9.81) | 69.1 (10.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 69 | 136
  Male | 37 | 32 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 32 | 40 | 72
  White | 68 | 57 | 125
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Age, Continous: Dose Maintenance Period [Mean (Standard Deviation); unit: years] — Population: Baseline data are reported for the Dose Maintenance Period, a subset of participants in the Safety Analysis Set starting the Dose Titration Period.
  years
    number analyzed (Participants) | 76 | 72 | 148
    (all) | 67.6 (11.57) | 69.6 (8.94) | 68.6 (10.38)
Sex: Female, Male: Dose Maintenance Period [Count of Participants; unit: Participants] — Population: Baseline data are reported for the Dose Maintenance Period, a subset of participants in the Safety Analysis Set starting the Dose Titration Period.
  Participants
    number analyzed (Participants) | 76 | 72 | 148
    Female | 46 | 48 | 94
    Male | 30 | 24 | 54
Race (NIH/OMB): Dose Maintenance Period [Count of Participants; unit: Participants] — Population: Baseline data are reported for the Dose Maintenance Period, a subset of participants in the Safety Analysis Set starting the Dose Titration Period.
  Participants
    number analyzed (Participants) | 76 | 72 | 148
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 26 | 29 | 55
    White | 48 | 40 | 88
    Unknown or Not Reported | 1 | 2 | 3
Hemoglobin [Mean (Standard Deviation); unit: grams per deciliter (g/dL)] — Population: Data are reported for Per-Protocol Analysis Set members, comprised of participants in the Full Analysis Set (FAS) (randomized participants who took >=1 dose of study medication and had >=1 post-randomization efficacy measurement) who met the study eligibility requirements and had no major protocol deviations that affected the validity of the efficacy measurements.
  grams per deciliter (g/dL)
    number analyzed (Participants) | 97 | 86 | 183
    (all) | 10.40 (0.749) | 10.51 (0.739) | 10.45 (0.744)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin (Hgb) at Week 24
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Estimates are from a mixed model of repeated measures (MMRM), including an intercept term and covariates for randomized treatment, visit, treatment by visit interaction, Baseline value, and Baseline value by visit interaction. The Kenward-Roger method was used along with an unstructured covariance matrix.
Time Frame: Baseline; Week 24
Population: Per-Protocol Analysis Set: participants in the Full Analysis Set (FAS) (randomized par. who took >=1 dose of study medication and had >=1 post-randomization efficacy measurement) who met the study eligibility requirements and had no major protocol deviations that affected the validity of the efficacy measurements. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: grams per deciliter (g/dL)
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 74 | 70
grams per deciliter (g/dL) | 0.73 (0.101) | 0.70 (0.104)

2. Secondary Outcome: Change From Baseline in Hgb at Week 48
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Estimates are from an MMRM, including an intercept term and covariates for randomized treatment, visit, treatment by visit interaction, Baseline value, and Baseline value by visit interaction. The Kenward-Roger method was used along with an unstructured covariance matrix.
Time Frame: Baseline; Week 48
Population: Per-Protocol Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 67 | 61
g/dL | 0.61 (0.114) | 0.58 (0.119)

3. Secondary Outcome: Time From Randomization to the First Increase From Baseline Hgb of at Least 0.5 Grams Per Deciliter (g/dL) During the Dose Titration Period
Description: The Kaplan-Meier estimator of the survival function of time from randomization to the first increase from Baseline Hgb of at least 0.5 g/dL for each of the two starting dose treatment groups were obtained.
Time Frame: from Randomization to Week 24
Population: Per-Protocol Analysis Set. Only participants with data available at Week 24 were analyzed. A participant's time to first hemoglobin value >= 0.5 above the Baseline value was censored at the study day of the participant's last hemoglobin assessment on or before the Week 24 visit.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 99 | 90
days | 84.0 [57.0 to 89.0] | 57.0 [29.0 to 85.0]

4. Secondary Outcome: Change From Baseline in Transferrin Saturation (TSAT) at Week 24
Description: as for outcome 2
Time Frame: Baseline; Week 24
Population: Per-Protocol Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percentage of transferrin saturation
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 75 | 69
percentage of transferrin saturation | 6.30 (1.023) | 6.85 (1.073)

5. Secondary Outcome: Change From Baseline in TSAT at Week 48
Description: as for outcome 2
Time Frame: Baseline; Week 48
Population: Per-Protocol Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percentage of transferrin saturation
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 68 | 61
percentage of transferrin saturation | 7.97 (1.053) | 10.63 (1.113)

6. Secondary Outcome: Change From Baseline in Ferritin at Week 24
Description: as for outcome 2
Time Frame: Baseline; Week 24
Population: Per-Protocol Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: nanograms per millilier (ng/mL)
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 75 | 70
nanograms per millilier (ng/mL) | 136.63 (13.315) | 155.28 (14.037)

7. Secondary Outcome: Change From Baseline in Ferritin at Week 48
Description: as for outcome 2
Time Frame: Baseline; Week 48
Population: Per-Protocol Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 69 | 62
ng/mL | 251.44 (29.417) | 343.27 (31.148)

8. Secondary Outcome: Change From Baseline in Serum Phosphate at Week 24
Description: as for outcome 2
Time Frame: Baseline; up to Week 24
Population: Per-Protocol Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 76 | 68
milligrams per deciliter (mg/dL) | -0.19 (0.065) | -0.25 (0.069)

9. Secondary Outcome: Change From Baseline in Serum Phosphate at Week 48
Description: as for outcome 2
Time Frame: Baseline; Week 48
Population: Per-Protocol Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 69 | 62
mg/dL | -0.07 (0.075) | -0.20 (0.079)

10. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 24
Description: as for outcome 2
Time Frame: Baseline; Week 24
Population: Per-Protocol Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: ml/minute/1.73 meters cubed (m^3)
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 76 | 68
ml/minute/1.73 meters cubed (m^3) | -1.08 (0.836) | -1.53 (0.0882)

11. Secondary Outcome: Change From Baseline in eGFR at Week 48
Description: as for outcome 2
Time Frame: Baseline; Week 48
Population: Per-Protocol Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: ml/minute/1.73 m^3
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 70 | 62
ml/minute/1.73 m^3 | -1.85 (0.977) | -2.20 (1.035)

12. Secondary Outcome: Change From Baseline in Bicarbonate at Week 24
Description: as for outcome 2
Time Frame: Baseline; Week 24
Population: Per-Protocol Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: milliquivalent (mEq)/Liter (L)
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 76 | 68
milliquivalent (mEq)/Liter (L) | -0.15 (0.296) | -0.05 (0.312)

13. Secondary Outcome: Change From Baseline in Bicarbonate at Week 48
Description: as for outcome 2
Time Frame: Baseline; Week 48
Population: Per-Protocol Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mEq/L
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 69 | 62
mEq/L | 0.03 (0.328) | -0.51 (0.345)

14. Secondary Outcome: Change From Baseline in Intact Parathyroid Hormone (iPTH) at Week 24
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Estimates obtained using a common slope analysis of covariance (ANCOVA) model which includes the Baseline laboratory parameter as a covariate, randomized treatment group, and a random error term.
Time Frame: Baseline; Week 24
Population: Per-Protocol Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: picograms per milliliter (pg/mL)
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 71 | 68
picograms per milliliter (pg/mL) | 1.64 (4.547) | 0.39 (4.647)

15. Secondary Outcome: Change From Baseline in iPTH at Week 48
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Estimates obtained using an uncommon slope ANCOVA model which includes the Baseline laboratory parameter as a covariate, randomized treatment group, randomized treatment group by Baseline interaction, and a random error term.
Time Frame: Baseline; Week 48
Population: Per-Protocol Analysis Set. Only participants who completed their Week 48 Visit were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 69 | 59
pg/mL | -1.49 (5.385) | 5.74 (5.824)

16. Secondary Outcome: Change From Baseline in C-terminal Fibroblast Growth Factor 23 (FGF23) at Week 24
Description: as for outcome 15
Time Frame: Baseline; Week 24
Population: Per-Protocol Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: relative units (RU)/mL
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 67 | 67
relative units (RU)/mL | -94.78 (26.393) | -63.22 (26.392)

17. Secondary Outcome: Change From Baseline in C-terminal FGF23 at Week 48
Description: as for outcome 15
Time Frame: Baseline; Week 48
Population: Per-Protocol Analysis Set. Only participants who completed their Week 48 Visit were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: RU/mL
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 65 | 58
RU/mL | -85.70 (23.029) | -80.34 (24.370)

18. Secondary Outcome: Change From Baseline in Intact Fibroblast Growth Factor 23 at Week 24
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Estimates obtained using a common slope ANCOVA model which includes the Baseline laboratory parameter as a covariate, randomized treatment group, and a random error term.
Time Frame: Baseline; Week 24
Population: Per-Protocol Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 70 | 67
pg/mL | -0.23 (8.106) | -2.01 (8.286)

19. Secondary Outcome: Change From Baseline in Intact Fibroblast Growth Factor 23 at Week 48
Description: as for outcome 15
Time Frame: Baseline; Week 48
Population: Per-Protocol Analysis Set. Only participants who completed their Week 48 Visit are included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 69 | 58
pg/mL | 18.52 (14.741) | 10.15 (16.086)

20. Secondary Outcome: Change From Baseline Scores for the Work Productivity and Activity Impairment (WPAI) Questionnaire Adapted for Anemia Associated With Chronic Kidney Disease (CKD) at Week 24: Work-associated Measures
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The WPAI is a questionnaire to evaluate the effect of anemia associated with Chronic Kidney Disease on the ability to work and perform regular activities. Scores are presented as percentages (multiplying the scores by 100), with 0% representing no impact and 100% representing complete impact.
Time Frame: Baseline; Week 24
Population: Per-Protocol Analysis Set. Only participants with available data who were currently employed (working for pay) were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of score
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 10 | 11
percentage of score
  Percent Work Time Missed: number analyzed (Participants) | 7 | 10
  Percent Work Time Missed | 0.00 (0.000) | -3.19 (9.222)
  Percent Impairment while Working: number analyzed (Participants) | 6 | 10
  Percent Impairment while Working | -15.00 (25.884) | 4.00 (30.258)
  Percent Overall Work Impairment: number analyzed (Participants) | 6 | 10
  Percent Overall Work Impairment | -15.00 (25.884) | 1.40 (26.842)

21. Secondary Outcome: Change From Baseline Scores for the WPAI Questionnaire Adapted for Anemia Associated With CKD at Week 48: Work-associated Measures
Description: as for outcome 20
Time Frame: Baseline; Week 48
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: percentage of score
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 14 | 11
percentage of score
  Percent Work Time Missed: number analyzed (Participants) | 7 | 9
  Percent Work Time Missed | 0.00 (0.000) | -3.48 (7.412)
  Percent Impairment while Working: number analyzed (Participants) | 7 | 9
  Percent Impairment while Working | -11.43 (16.762) | 7.78 (29.486)
  Percent Overall Work Impairment: number analyzed (Participants) | 7 | 9
  Percent Overall Work Impairment | -11.43 (16.762) | 4.71 (24.601)

22. Secondary Outcome: Change From Baseline Scores for the WPAI Questionnaire Adapted for Anemia Associated With CKD at Week 24: Activity Impairment
Description: as for outcome 20
Time Frame: Baseline; Week 24
Population: Per-Protocol Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of score
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 76 | 71
percentage of score | -18.03 (28.753) | -6.34 (31.769)

23. Secondary Outcome: Change From Baseline Scores for the WPAI Questionnaire Adapted for Anemia Associated With CKD at Week 48: Activity Impairment
Description: as for outcome 20
Time Frame: Baseline; Week 48
Population: Per-Protocol Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of score
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 70 | 61
percentage of score | -16.71 (36.859) | -6.72 (36.227)

24. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale Score at Week 24
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Participants were asked to respond to 13 statements (as they apply to the last 7 days) that other people with the same illness said are important with one of the following: 0, not at all; 1, a little bit; 2, somewhat; 3, quite a bit; 4, very much. All individual items were summed to create a single fatigue score ranging from 0 to 52. Higher scores indicate greater fatigue.
Time Frame: Baseline; Week 24
Population: Per-Protocol Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 77 | 72
score on a scale | 7.22 (10.986) | 4.35 (10.047)

25. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy Fatigue Scale Score at Week 48
Description: as for outcome 24
Time Frame: Baseline; Week 48
Population: Per-Protocol Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 69 | 62
score on a scale | 7.49 (11.817) | 3.68 (9.954)

26. Secondary Outcome: Number of Hospitalizations for Participants Who Entered the Dose Maintenance Period
Description: A hospitalization is defined as admission to the hospital.
Time Frame: up to Week 48
Population: Per-Protocol Analysis Set
Measure: Number; unit: hospitalizations
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 97 | 86
hospitalizations | 13 | 10

27. Secondary Outcome: Duration of Hospitalizations for Participants Who Entered the Dose Maintenance Period
Description: A hospitalization is defined as admission to the hospital.
Time Frame: up to Week 48
Population: Per-Protocol Analysis Set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 13 | 10
days | 4.08 (2.499) | 3.91 (0.980)

28. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE) for Participants Who Entered the Dose Maintenance Period
Description: Treatment-emergent adverse events are defined as adverse events that began after the first administration of study medication or pre-existing conditions that worsened after the first dose of study medication.
Time Frame: up to Week 48
Population: Safety Analysis Set: all participants who took at least 1 dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
Number analyzed (Participants) | 104 | 101
Participants | 89 | 89

ADVERSE EVENTS:
Time Frame: from the time of informed consent up to 48 weeks
Description: Treatment-emergent adverse events, defined as adverse events that began after the first administration of study medication or pre-existing conditions that worsened after the first dose of study medication, were collected in members of the Safety Analysis Set (comprised as all participants who took at least 1 dose of study medication). Data are reported for those participants who entered the Dose Maintenance Period.
Arm/Group | KRX-0502 3 g/Day | KRX-0502 4 g/Day
All-Cause Mortality (participants affected / at risk) | 3/104 | 2/101
Serious Adverse Events (participants affected / at risk) | 26/104 | 25/101
Other Adverse Events (participants affected / at risk) | 58/104 | 59/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KRX-0502 3 g/Day (N=104) | KRX-0502 4 g/Day (N=101)
Cellulitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Chest wall abscess (Infections and infestations) | 1 | 0
Cystitis escherichia (Infections and infestations) | 1 | 0
Enterobacter sepsis (Infections and infestations) | 0 | 1
Escherichia pyelonephritis (Infections and infestations) | 1 | 0
Gastritis viral (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Infectious colitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Viral sepsis (Infections and infestations) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 4
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Internal hernia (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 5
End stage renal disease (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Malignant hypertension (Vascular disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Ureteric injury (Injury, poisoning and procedural complications) | 0 | 1
Brain stem stroke (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Anticoagulation drug level above therapeutic (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | KRX-0502 3 g/Day (N=104) | KRX-0502 4 g/Day (N=101)
Constipation (Gastrointestinal disorders) | 17 | 12
Diarrhoea (Gastrointestinal disorders) | 13 | 15
Faeces discoloured (Gastrointestinal disorders) | 16 | 10
Urinary tract infection (Infections and infestations) | 15 | 11
Hypertension (Vascular disorders) | 12 | 11
Nausea (Gastrointestinal disorders) | 8 | 11
Oedema peripheral (General disorders) | 5 | 9
Vomiting (Gastrointestinal disorders) | 2 | 8
Dizziness (Nervous system disorders) | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT03236246/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT03236246/SAP_001.pdf